CLINICAL TRIAL: NCT03172923
Title: Randomised Trial of Trochanteric Hip Fractures Treated With Either a Sliding Hip Screw on an Intramedullary Nail
Brief Title: Nail Versus Sliding Hip Screw for Trochanteric Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peterborough and Stamford Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Martyn J Parker, Consultant orthopaedic surgeon, Peterborough and Stamford Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC 10/H0306/66
Record Dates: First submitted 2017-05-26; First posted 2017-06-01 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: outcome assessor is blinded to treatment given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sliding hip screw (Active Comparator): fixation of fracture with a sliding hip screw
  Interventions: Device: sliding hip screw
- intramedullary nail (Experimental): fixation of the fracture with an intramedullary nail
  Interventions: Device: intramedullary nial

INTERVENTIONS:
Device: sliding hip screw — fixation of the fracture with a sliding hip screw
  Arms: sliding hip screw
Device: intramedullary nial — fixation of the fracture with an intramedullary nail
  Arms: intramedullary nail

SUMMARY:
The investigators therefore propose to undertake a further randomised controlled trial comparing the sliding hip screw (SHS) with the Targon PFT intramedullary nail. The aim is to see if the summation of the first trial of 600 participants comparing the sliding hip screw with the Targon PF nails, in conjunction with this study of 400 participants with the updated Targon PFT nail produces results that convincingly demonstrate that this particular design of implant is superior to the sliding hip screw. Because of the financial issues involved a cost benefit comparison for the two procedures is planned at the completion of the study.

Primary outcome measures will be regain of walking ability. Secondary outcome measures recorded with include mortality, length of surgery, operative blood loss, blood transfusion, post-operative complications, hospital stay, need for subsequent revision surgery and degree of residual pain.

DETAILED DESCRIPTION:
The trial will be run as close to the ideal trial methodology for a randomised trial as specified by the CONSORT statement as possible. This will include secure randomisation, intention to treat analysis, full reporting of outcomes and follow-up by a person who is blinded to the prosthesis used. The trial will follow the code of good clinical practice as specified by the hospital trusts Research and Development Committee.

In Peterborough all hip fracture patients are admitted to the acute trauma ward and transferred to the care of MJP. Those patients that are willing to participant in one of our randomised trials are consented prior to surgery. Treatment follows standard evidence based protocols with follow-up of all patients in a hip fracture clinic. A comprehensive database is maintained for all patients containing both audit and research data. Included in this is a standardised assessment of outcome.

The sliding hip screw used if of a standard design that has been in use at Peterborough for the last fifty years. The intramedullary nails used will be the Targon PFT nail. This nail is very similar to the Targon PF nail used in the earlier trial on this topic. Bases on the results of the previous study and the experience of other users the nail has undergone minor modifications that are primarily aimed at making the nail easier to use with improved instrumentation and also a change to design of the cross screw aimed at reducing the risk of fracture fixation complications occurring.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Peterborough District Hospital with a trochanteric hip fracture that is to be treated by internal fixation.

Exclusion Criteria:

* Patients who decline to participate
* Patients without the capacity to give informed consent
* Patients admitted when MJP is not available to supervise treatment
* Patients with pathological fractures from Paget's disease of bone secondaries from tumour

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-10-08 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
regain of mobility | one year from injury
  regain of walking ability using a standardised mobility score (Parker MJ, Palmer CR. A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg 1993;75-B:797-8.)

SECONDARY OUTCOMES:
mortality | at one year from injury
  mortality

IPD SHARING:
Plan to Share IPD: No